CLINICAL TRIAL: NCT06552962
Title: Effects of Whole Body Vibration on Pain, Function and Viscoelasticity in Patients With Non-Specific Low Back Pain
Brief Title: Effects of Whole Body Vibrationin in Patients With Non-Specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Collaborators: Istinye University (Other)
Responsible Party: Principal Investigator, Beyza Tanrıöğen, Research Assistant (MSc student), Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: İÜC-BT1
Record Dates: First submitted 2024-07-25; First posted 2024-08-14 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Low Back Pain; Low Back Pain, Mechanical; Low Back Pain, Postural; Low Back Pain, Recurrent
Keywords: whole body vibration; biomechanical structures; low back pain; core stabilisation; lumbar myofascia
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Within the scope of the research, individuals with chronic non-specific low back pain will be randomized and divided into two separate groups. The control group will undergo lumbar stabilization exercises twice a week for 6 weeks. The experimental group will have the same lumbar stabilization exercises performed on the whole body vibration device twice a week for 6 weeks. The frequency of the device will be set to 30 Hz. Exercise duration, frequency, number and variety will be kept equal for the experimental and control groups. Demographic information of the patients, viscoelastic properties of the lumbar region, pain, function, quality of life, lower extremity muscle strength, endurance, balance and proprioception will be evaluated. Measurements will be made before treatment and at the end of 6 weeks of treatment.
Who Masked: Participant, Outcomes Assessor
Masking Description: The study was designed as a double-blind randomize-controlled study in which the participant and the evaluator were blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The experimental group will have the same lumbar stabilization exercises performed on the whole body vibration device twice a week for 6 weeks. The frequency of the device will be set to 30 Hz. Exercise duration, frequency, number and variety will be kept equal for the experimental and control groups. Demographic information of the patients, viscoelastic properties of the lumbar region, pain, function, quality of life, lower extremity muscle strength, endurance, balance and proprioception will be evaluated. Measurements will be made before treatment and at the end of 6 weeks of treatment.
  Interventions: Device: Whole body vibration
- Control Group (Active Comparator): Within the scope of the research, individuals with chronic non-specific low back pain will be randomized and divided into two separate groups. Lumbar stabilization exercises will be applied to the control group twice a week for 6 weeks. Exercise duration, frequency, number and variety will be kept equal for the experimental and control groups. Demographic information of the patients, viscoelastic properties of the lumbar region, pain, function, quality of life, lower extremity muscle strength, endurance, balance and proprioception will be evaluated. Measurements will be made before treatment and at the end of 6 weeks of treatment.
  Interventions: Behavioral: lumbar stabilization exercises

INTERVENTIONS:
Device: Whole body vibration — The aim of this study is to reveal the effect of exercises performed with WBV on the myofascial tissue of the lumbar region and the tone of superficial back muscles, as well as to investigate the effects on pain, function, muscle strength, balance, proprioception and endurance parameters, compared to the exercise-only group.
  Arms: Intervention Group
Behavioral: lumbar stabilization exercises — The control group will undergo lumbar stabilization exercises twice a week for 6 weeks.
  Arms: Control Group

SUMMARY:
After acute low back pain, one third of patients have chronic low back pain. A sedentary lifestyle is a leading cause of mechanical stress-related low back pain and exacerbates chronic low back pain. Balance disorders, postural adjustment disorder, abnormal spinal movements and related muscle imbalance are observed in individuals with chronic low back pain. Conservative treatment is mostly used in treatment. Langevin et al. stated that an abnormal and irregular thoracolumbar connective tissue structure is observed in chronic and recurrent low back pain. It has been said that physiotherapy and rehabilitation methods such as exercise therapy, massage, chiropractic and acupuncture provide changes in the biomechanical components of the affected connective tissue such as stiffness, viscoelasticity and density. Over the past 20 years, exercises with Whole Body Vibration (WBV) have begun to be used as an effective method for reducing pain. Exercises performed with WBV are thought to improve neuromuscular activation and increase muscle strength and joint stabilization. In non-specific chronic low back pain, increased tone is observed in the superficial back muscles. And based on this study, no study has been found examining the effect of vibratory exercise intervention on the tone of superficial back muscles that go into spasm due to pain. In this study, lumbar stabilization exercises, one of the most effective exercise methods in chronic low back pain, will be applied and exercises performed with vibration will have an additional effect.

It is aimed to reveal whether it creates or not. MyotonPRO (myometer) is a digital palpation device that can measure the viscoelastic properties of myofascial tissue. In measurements made with patients with chronic low back pain and healthy controls, While lumbar myofascial tissue elasticity was significantly low in patients; The tone of the lumbar extensor muscles was found to be significantly higher. However, this measurement has not been made before in studies conducted with WBV, which is one of the methods used to reduce pain in individuals with chronic low back pain.

The aim of this study is to reveal the effect of exercises performed with WBV on the myofascial tissue of the lumbar region and the tone of the superficial back muscles, on pain, function, muscle strength, balance, proprioception and endurance parameters compared to the group exercising only.

DETAILED DESCRIPTION:
WBV exercise is a popular method to reduce pain intensity and improve function and quality of life.

is the method. WBV exercise is currently used as a treatment for patients with chronic low back pain. The effect of WBV exercise on the treatment of low back pain can be explained by activating the core muscles and increasing stabilization. Additionally, paravertebral muscle spasm occurs in most patients, and it is said that WBV can relieve pain by relaxing the paravertebral muscles. In addition, it is thought that it may reduce the associated spinal dysfunction and instability by improving the proprioception of the lumbosacral region. Although studies have begun with WBV in patient groups with chronic low back pain, the studies are limited.

Therefore, the optimal dosage has not yet been determined. It aims to compare its effect on strength, balance, proprioception, endurance, quality of life and viscoelastic properties of the lumbar region. Thus, WBV on the specified parameters It is aimed to reveal its effectiveness and contribute to the existing literature. Measurement with the MyotonPRO device, a newly widespread and expensive measuring device, will strengthen the objective and original aspect of the study. Lumbar stabilization exercises (LSE) try to correct the disorders by activating the trunk muscles. In this respect, it is widely used by physiotherapists in the treatment of low back pain. In our study, while lumbar stabilization exercises were applied to individuals in the control group; intervention The group will be given exercise accompanied by vibration. The effect of the added vibration on the exercises accepted in the literature will be examined. The effectiveness of WBV in patients with chronic non-specific low back pain will be evaluated by making the following measurements: MyotonPRO: The measurement will be made in the prone position, without active muscle contraction. Lumbar paraspinal muscle measurement will be made from a point one finger to the right/left of the L4 level.

Pain: Participants' pain intensity will be evaluated according to the Visual Analog Scale (VAS).

Function: The Oswestry Low Back Pain Disability Questionnaire measures the functioning of patients affected by low back pain.

It is an index consisting of 10 sections used for evaluation. Quality of Life: Measurement with Short Form SF-12, which is the abbreviated version of the SF-36 Quality of Life Scale will be done. Lower Extremity Muscle Strength: Myometer is a muscle strength measurement device. More objective than manual muscle testing provides data. Endurance: The endurance of the trunk muscles is measured by lateral bridging, Sorensen and trunk flexors endurance test.

will be measured. Balance: Dynamic balance will be measured with the Y balance test. Static Balance, Single Leg Stand Test will be done. This test is performed with eyes open and hands on hips. Proprioception: With the passive positioning technique, a certain angle is applied to the lumbar region as the patient's eyes are closed.

Position is given passively with the helper and then the patient is asked to do the same without support using the same extremity.

You are asked to find the angle. The difference between the angles is recorded with a goniometer.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with Non-Specific low back pain by a physician,
* Having a complaint of non-specific low back pain for at least 3 months,
* Being 18 years or older,
* Volunteer,
* Not having any diagnosed cardiac disease,
* Not having any diagnosed neuromuscular disease,
* Pain level should be at least 3 according to VAS,
* Not having received physiotherapy or rehabilitation in the last 3 months
* Individuals who meet the above criteria will be included in the study.

Exclusion Criteria:

* Diagnosed stomach, kidney, liver, pancreas and bladder problems,
* Presence of mental or cognitive problems,
* History of surgery for low back pain,
* Pain level is 8 or above according to Visual Analogue Scale,
* Use of painkillers during treatment,
* Acute and severe musculoskeletal pain,
* Radiculopathy,
* Malignancy,
* Pregnancy,
* Pace maker users,
* Epilepsy,

Individuals meeting the above criteria will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2024-07-25 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2025-02-06 (Actual)

PRIMARY OUTCOMES:
MyotonPRO myofascial palpation device | 6 weeks
  The measurement will be made in the prone position, without active muscle contraction. Lumbar paraspinal muscle measurement will be made from a point one finger to the right/left of the L4 level.
  F - Natural Oscillation Frequency [Hz], characterizing Tone or Tension S - Dynamic Stiffness [N/m] D - Logarithmic Decrement [relative unit], characterizing Elasticity R - Mechanical Stress Relaxation Time [ms] C - Ratio of Relaxation and Deformation time [relative unit], characterizing Creep

SECONDARY OUTCOMES:
Pain severity for lower back (Visual analog scale) | 6 weeks
  Participants' pain intensity will be evaluated according to Visual Analog Scale. The score is from 0 to 10. The pain level increases from 0 to 10.
Low Back Function Assesment | 6 weeks
  The Oswestry Low Back Pain Disability Questionnaire is a 10-part index used to assess the functioning of patients affected by low back pain.
Quality of Life (SF-12 SHORT FORM) | 6 weeks
  Measurement will be made with Short Form SF-12, which is the shortened version of the SF-36 Quality of Life Scale.
Lower Extremity Muscle Strength | 6 weeks
  Myometer is a muscle strength measurement device. Provides more objective data than manual muscle testing.
Abdominals, side abdominals and back extenstors Endurance | 6 weeks
  The endurance of the trunk muscles will be measured by lateral bridging, Sorensen and trunk flexors endurance test.
Dynamic Balance | 6 weeks
  Dynamic balance will be measured with the Y balance test.
Lumbar Proprioception | 6 weeks
  With the passive positioning technique, a certain angle is applied to the lumbar region with the patient's eyes closed.
  The position is given passively and then the patient is asked to find the same angle without support, using the same extremity. The difference between the angles is recorded with a goniometer [29]
Static Balance | 6 weeks
  Static Balance and Single Leg Standing Test will be performed. This test is performed with eyes open and hands on hips.

CONTACTS AND LOCATIONS:
Overall Officials: Yıldız Analay Akbaba, Phd, Study Director — Istanbul University - Cerrahpasa; Beyza Tanrıöğen, MSc (c), Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istinye University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No